CLINICAL TRIAL: NCT05336851
Title: Emergency PanorOmic Wide Association Study in Respiratory Infectious Disease (ePWAS-RID)
Brief Title: Emergency PWAS in Respiratory Infectious Disease
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Timothy Hudson RAINER, Professor of Department of Emergency Medicine, The University of Hong Kong
Other Study IDs: ePWAS-RID/Rainer/2021
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Viral Infections; Bacterial Infections; Fungal Infections; Mixed Infection; Mycobacterium Infection; Infection of Uncertain Aetiology; Pneumonia; Sepsis
Keywords: Biobank; Diagnostics and Prognostics; Emergency Medicine; Multiomics and Panoromics; Respiratory Infectious Disease
MeSH Terms: conditions — Virus Diseases; Bacterial Infections; Mycoses; Coinfection; Mycobacterium Infections; Pneumonia; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — At least one whole blood and saliva drawn a) in the emergency department (if available) or hospital within 8 days of the onset of symptoms; and if they agree, a further two samples at b) 24 hours +/- 6 hours from symptom onset (if available); and c) 48 hours +/- 6 hours from symptom onset (if available).
  Liquid biopsy for retention:
  • Whole Blood samples, red blood cell effluent, plasma, white cell pellet(for genomic, epigenomic, transcriptomic and proteomic studies). serum (for proteomic, metabolomic and lipidomic studies), salivary supernatant, salivary cells. Biomarkers under investigation: DNA gene expression, RNA gene expression, Proteomics expression, Metabolomics expression and Lipidomics expression in peripheral blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Viral infection: Viral infection subjects presenting within 8 days from symptom onset will have at least one whole blood and saliva drawn a) in the emergency department (if available) or hospital within 8 days of the onset of symptoms; and if they agree
  Interventions: Diagnostic Test: Biomarker blood draw and saliva collection
- Bacterial infection: Bacterial infection subjects presenting within 8 days from symptom onset will have at least one whole blood and saliva drawn a) in the emergency department (if available) or hospital within 8 days of the onset of symptoms; and if they agree, a further two samples at b) 24 hours +/- 6 hours from symptom onset (if available); and c) 48 hours +/- 6 hours from symptom onset (if available).
  Interventions: Diagnostic Test: Biomarker blood draw and saliva collection
- Viral-Viral co-infection: Viral-viral co-infection subjects presenting within 8 days from symptom onset will have at least one whole blood and saliva drawn a) in the emergency department (if available) or hospital within 8 days of the onset of symptoms; and if they agree, a further two samples at b) 24 hours +/- 6 hours from symptom onset (if available); and c) 48 hours +/- 6 hours from symptom onset (if available).
  Interventions: Diagnostic Test: Biomarker blood draw and saliva collection
- Bacterial-Viral co-infection: Bacterial-Viral co-infection subjects presenting within 8 days from symptom onset will have at least one whole blood and saliva drawn a) in the emergency department (if available) or hospital within 8 days of the onset of symptoms; and if they agree, a further two samples at b) 24 hours +/- 6 hours from symptom onset (if available); and c) 48 hours +/- 6 hours from symptom onset (if available).
  Interventions: Diagnostic Test: Biomarker blood draw and saliva collection
- Fungal-Mycobacterium co-infection: Bacterial-Viral co-infection subjects presenting within 8 days from symptom onset will have at least one whole blood and saliva drawn a) in the emergency department (if available) or hospital within 8 days of the onset of symptoms; and if they agree, a further two samples at b) 24 hours +/- 6 hours from symptom onset (if available); and c) 48 hours +/- 6 hours from symptom onset (if available).
  Interventions: Diagnostic Test: Biomarker blood draw and saliva collection
- Infection of uncertain origin: Infection of uncertain origin subjects presenting within 8 days from symptom onset will have at least one whole blood and saliva drawn a) in the emergency department (if available) or hospital within 8 days of the onset of symptoms; and if they agree, a further two samples at b) 24 hours +/- 6 hours from symptom onset (if available); and c) 48 hours +/- 6 hours from symptom onset (if available).
  Interventions: Diagnostic Test: Biomarker blood draw and saliva collection
- Control Subjects: Control group subjects, if they agree, will have at least one whole blood and saliva drawn a) in the emergency department (if available) or hospital within 8 days of the onset of symptoms (if applicable); and if they agree, a further two samples at b) 24 hours +/- 6 hours from symptom onset (if applicable); and c) 48 hours +/- 6 hours from symptom onset (if applicable).
  Interventions: Diagnostic Test: Biomarker blood draw and saliva collection

INTERVENTIONS:
Diagnostic Test: Biomarker blood draw and saliva collection — Three peripheral 10 - 20mL blood sample (if available) Three 1 - 5mL salivary samples (if available)

SUMMARY:
Develop an emergency PanorOmics Wide Association Study (ePWAS) for the early, rapid biological and pathophysiological characterisation of known and novel Infectious Diseases in adult patients presenting to emergency departments with suspected, acute, community-acquired respiratory infectious disease (scaRID).

Phase 1

1. Develop an ED-ID biobank (named ePWAS-RID). Phase 2
2. Targeted research for the discovery of novel diagnostics, prognostics and therapeutics

DETAILED DESCRIPTION:
Introduction

Pandemic Preparedness

The COVID-19 pandemic has affected over 220 million people, claimed over 450 000 lives and invoked variable responses across the world. Delays in acquiring quality clinical and scientific material on the transmissibility, clinical nature, outcomes and lethality of novel and known infectious diseases (ID) translate into healthcare inefficiencies, societal and economic stress, and increased morbidity and mortality. Regions with greater success in the fight against COVID-19 were well prepared before the pandemic.

Pathogens

The pathogens most likely to cause annual epidemics and pandemics are respiratory viruses. In Asia, viral infections account for 30-40% of sepsis cases. Each year there are 100 million cases of viral community-acquired pneumonia (CAP) of which 60% progress to sepsis. These viruses cause host-mediated, inflammatory, immune responses which progresses through three phases: preliminary regulated inflammation; intermediate dysregulated proinflammation; and late dysregulated hypoinflammation.

Clinical Spectrum

RID is a heterogeneous population of patients. This complex spectrum of heterogeneity extends throughout the underlying molecular biology and pathophysiology from genome to phenome. It includes significant individual variation in regulated and dysregulated systemic inflammatory host responses to infection in the presence and absence of organ dysfunction. Critical illness from any ID involves both host susceptibility to the pathogen and host propensity to develop dysregulated inflammation and organ failure (e.g. pulmonary inflammation and/or acute kidney injury).

PanorOmics-Wide Association Studies

In the five years prior to the COVID-19 pandemic, the United Kingdom's Genetics Of Mortality In Critical Care (GenOMICC) study recruited patients with a spectrum of critical illness syndromes (e.g. influenza, sepsis, and emerging infections) to better understand host mechanisms that lead to life-threatening outcomes. As a result, the GenOMICC investigators, along with collaborators from Spain and Italy, were well placed to perform genomic-association studies on critically ill COVID-19 patients and to make recommendations for future studies.

An integrated panorOmics approach has the potential to uncover causal associations and linkages across the entire spectrum of host biology including genomics, epigenomics, transcriptomics, proteomics, metabolomics and lipidomics, through to clinical phenotype. However, panorOmics as a discipline faces the same challenges as Genome-wide association studies (GWAS), only more so. Although GWAS correlate genomic loci with complex signatures and traits, efficient detection is hindered by false positives, linkage disequilibrium, and high expense. True causal variations and real underlying associations require multiple filters if they are to be detected.

The investigators propose to develop an ED-based system of dynamic studies on blood and saliva samples taken from patients at an early stage of ID. Early stage refers to a process in the patient pathway that precedes most patient recruitment in other studies i.e. on wards or ICU. The two primary objectives are a) to develop an ED-ID biobank; and b) to undertake preliminary discovery and targeted research for the discovery of novel diagnostics, prognostics and therapeutics.

The investigators will define early multiOmics signatures of RID and identify relationships to known and novel ID. Few studies have been published on the integrated panorOmics of COVID-19, and few if any address the early phases of illness or differentiating features in comparison to other respiratory illnesses.

In disease stratified, case-control matched comparisons of adult patients with scaRID attending EDs, what panorOmic signatures differentiate low risk from high risk across a 30-day WHO-Clinical Progression Scale (WHO-CPS)?

For the purpose of this study, scaRID is defined as:

1. A fever or a temperature >37.5°C; AND
2. One or more relevant symptoms:

   * respiratory symptoms (e.g. cough, shortness of breath), OR
   * systemic symptoms (e.g. chills, rigors, myalgia), OR
   * gastrointestinal symptoms (e.g. nausea, vomiting, diarrhoea); AND
3. No obvious alternative cause (see exclusion criteria).

PanorOmic associations will be derived from liquid biopsy samples, including whole blood, plasma, serum, white cell pellet, red cell effluent, salivary supernatant, and salivary cells. Liquid biopsy biomarkers include genomic, transcriptomic, proteomic, metabolomic, lipidomic and haematological contents.

Hypothesis The investigators hypothesise that in propensity-matched, adult patients with pathogen-specific and disease specific RID (e.g. SARS-CoV-2, Influenza A) there are significant differences in panorOmic signatures that delineate host susceptibility and host response for mild to severe disease.

Objectives

The purpose of this proposal is to develop an emergency PanorOmics Wide Association Study (ePWAS) biobank for the early, rapid biological and pathophysiological characterisation of scaRID. More specifically, in adult patients presenting to EDs with scaRID and within 10 days of symptom onset, we aim:

1. To develop an ED-ePWAS-RID biobank of blood and saliva samples
2. To use this databank for exploratory and targeted research in the search for diagnostic and prognostic markers and to understand underlying mechanisms of disease

The goals of the biobank and the ePWAS-RID repository are:

* to develop the infrastructure for a sustainable ED-based biobank of blood and saliva samples matched to clinical phenotypes and critical outcomes.
* to develop the repository according to international standards thereby minimising heterogeneity and rendering the material suitable for international research frameworks that aims to facilitate access to human biological materials.
* to prepare a repository for preliminary discovery of novel diagnostic, prognostic, and therapeutic markers.
* to facilitate targeted research on the pathogenesis of respiratory infections, host susceptibility, and host response.
* to derive biomarker platforms of training set models for early RID detection, pathogen differentiation, monitoring, risk stratification and prognosis; and to validate those models using independent and external datasets.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for enrolment include:

With reference to previous inclusion criteria are:

* Adults ≥18 years of age; AND
* Suspected, acute, community-acquired, respiratory, infectious disease (scaRID)*; AND
* Informed consent.

Note: scaRID is defined according to ALL three criteria:

1. Community acquired (not hospitalised for <28 days); AND
2. Acute infection (defined as symptom onset <8 days and any ONE of reported fever or chills or aural temperature >37.5°C or hypothermia or leucocytosis or leucopaenia or new altered mental status); AND
3. Probable respiratory infection - According to any ONE of:

   1. new cough or new sputum production or
   2. chest pain or
   3. dyspnoea or
   4. tachypnoea or
   5. abnormal lung examination or
   6. respiratory failure; or
   7. physician's judgment (presenting with systemic or gastrointestinal symptoms).

Control subjects will be drawn from two groups:

* The worried well - adult patients with a National Early Warning Score (NEWS) <3 and a temperature <37.5°C.
* Relatives or accompanying friends with no acute illness.

Exclusion Criteria:

* Refusal of consent;
* Recent hospitalisation (<28 days);
* Enrolled in another clinical trial
* Cellulitis;
* Skin or orthopaedic infections;
* Urinary tract infection;
* Acute abdominal sepsis;
* Sexual transmitted disease;
* Human immunodeficiency virus (HIV) infection;
* Immunocompromised/potential neutropenic fever;
* Solid organ or haematopoietic stem-cell transplant within the previous 90 days;
* Active graft-versus-host disease or bronchiolitis obliterans;
* Severe traveller's disease requiring urgent hospitalisation and management including malaria, dengue, typhoid and other rickettsial diseases;
* Stroke;
* Toxidrome;
* Non-organic acute psychosis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Suspected, acute, community-acquired, respiratory, infectious disease presenting to emergency department with symptom onset <8 days and reported fever or chills or aural temperature >37.5°C
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
WHO-CPS | Up to 30 days
  Differentiation of WHO-CPS >6 from WHO-CPS ≤6

SECONDARY OUTCOMES:
Mortality | Up to 30 days
  Mortality is defined as all-cause, Binary: Yes or No
Mortality | one year
  Mortality is defined as all-cause, Binary: Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H Rainer, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharfstein JM, Becker SJ, Mello MM. Diagnostic Testing for the Novel Coronavirus. JAMA. 2020 Apr 21;323(15):1437-1438. doi: 10.1001/jama.2020.3864. No abstract available. PMID 32150622
- [Background] Leung K, Wu JT, Liu D, Leung GM. First-wave COVID-19 transmissibility and severity in China outside Hubei after control measures, and second-wave scenario planning: a modelling impact assessment. Lancet. 2020 Apr 25;395(10233):1382-1393. doi: 10.1016/S0140-6736(20)30746-7. Epub 2020 Apr 8. PMID 32277878
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] He X, Lau EHY, Wu P, Deng X, Wang J, Hao X, Lau YC, Wong JY, Guan Y, Tan X, Mo X, Chen Y, Liao B, Chen W, Hu F, Zhang Q, Zhong M, Wu Y, Zhao L, Zhang F, Cowling BJ, Li F, Leung GM. Temporal dynamics in viral shedding and transmissibility of COVID-19. Nat Med. 2020 May;26(5):672-675. doi: 10.1038/s41591-020-0869-5. Epub 2020 Apr 15. PMID 32296168
- [Background] Williamson EJ, Walker AJ, Bhaskaran K, Bacon S, Bates C, Morton CE, Curtis HJ, Mehrkar A, Evans D, Inglesby P, Cockburn J, McDonald HI, MacKenna B, Tomlinson L, Douglas IJ, Rentsch CT, Mathur R, Wong AYS, Grieve R, Harrison D, Forbes H, Schultze A, Croker R, Parry J, Hester F, Harper S, Perera R, Evans SJW, Smeeth L, Goldacre B. Factors associated with COVID-19-related death using OpenSAFELY. Nature. 2020 Aug;584(7821):430-436. doi: 10.1038/s41586-020-2521-4. Epub 2020 Jul 8. PMID 32640463
- [Background] Pairo-Castineira E, Clohisey S, Klaric L, Bretherick AD, Rawlik K, Pasko D, Walker S, Parkinson N, Fourman MH, Russell CD, Furniss J, Richmond A, Gountouna E, Wrobel N, Harrison D, Wang B, Wu Y, Meynert A, Griffiths F, Oosthuyzen W, Kousathanas A, Moutsianas L, Yang Z, Zhai R, Zheng C, Grimes G, Beale R, Millar J, Shih B, Keating S, Zechner M, Haley C, Porteous DJ, Hayward C, Yang J, Knight J, Summers C, Shankar-Hari M, Klenerman P, Turtle L, Ho A, Moore SC, Hinds C, Horby P, Nichol A, Maslove D, Ling L, McAuley D, Montgomery H, Walsh T, Pereira AC, Renieri A; GenOMICC Investigators; ISARIC4C Investigators; COVID-19 Human Genetics Initiative; 23andMe Investigators; BRACOVID Investigators; Gen-COVID Investigators; Shen X, Ponting CP, Fawkes A, Tenesa A, Caulfield M, Scott R, Rowan K, Murphy L, Openshaw PJM, Semple MG, Law A, Vitart V, Wilson JF, Baillie JK. Genetic mechanisms of critical illness in COVID-19. Nature. 2021 Mar;591(7848):92-98. doi: 10.1038/s41586-020-03065-y. Epub 2020 Dec 11. PMID 33307546
- [Background] Legido-Quigley H, Asgari N, Teo YY, Leung GM, Oshitani H, Fukuda K, Cook AR, Hsu LY, Shibuya K, Heymann D. Are high-performing health systems resilient against the COVID-19 epidemic? Lancet. 2020 Mar 14;395(10227):848-850. doi: 10.1016/S0140-6736(20)30551-1. Epub 2020 Mar 6. No abstract available. PMID 32151326
- [Background] Lam TT, Jia N, Zhang YW, Shum MH, Jiang JF, Zhu HC, Tong YG, Shi YX, Ni XB, Liao YS, Li WJ, Jiang BG, Wei W, Yuan TT, Zheng K, Cui XM, Li J, Pei GQ, Qiang X, Cheung WY, Li LF, Sun FF, Qin S, Huang JC, Leung GM, Holmes EC, Hu YL, Guan Y, Cao WC. Identifying SARS-CoV-2-related coronaviruses in Malayan pangolins. Nature. 2020 Jul;583(7815):282-285. doi: 10.1038/s41586-020-2169-0. Epub 2020 Mar 26. PMID 32218527
- [Background] Hung IF, Lung KC, Tso EY, Liu R, Chung TW, Chu MY, Ng YY, Lo J, Chan J, Tam AR, Shum HP, Chan V, Wu AK, Sin KM, Leung WS, Law WL, Lung DC, Sin S, Yeung P, Yip CC, Zhang RR, Fung AY, Yan EY, Leung KH, Ip JD, Chu AW, Chan WM, Ng AC, Lee R, Fung K, Yeung A, Wu TC, Chan JW, Yan WW, Chan WM, Chan JF, Lie AK, Tsang OT, Cheng VC, Que TL, Lau CS, Chan KH, To KK, Yuen KY. Triple combination of interferon beta-1b, lopinavir-ritonavir, and ribavirin in the treatment of patients admitted to hospital with COVID-19: an open-label, randomised, phase 2 trial. Lancet. 2020 May 30;395(10238):1695-1704. doi: 10.1016/S0140-6736(20)31042-4. Epub 2020 May 10. PMID 32401715
- [Background] Tsang KW, Ho PL, Ooi GC, Yee WK, Wang T, Chan-Yeung M, Lam WK, Seto WH, Yam LY, Cheung TM, Wong PC, Lam B, Ip MS, Chan J, Yuen KY, Lai KN. A cluster of cases of severe acute respiratory syndrome in Hong Kong. N Engl J Med. 2003 May 15;348(20):1977-85. doi: 10.1056/NEJMoa030666. Epub 2003 Mar 31. PMID 12671062
- [Background] Wai AKC, Wong CKH, Wong JYH, Xiong X, Chu OCK, Wong MS, Tsui MSH, Rainer TH. Changes in Emergency Department Visits, Diagnostic Groups, and 28-Day Mortality Associated With the COVID-19 Pandemic: A Territory-Wide, Retrospective, Cohort Study. Ann Emerg Med. 2022 Feb;79(2):148-157. doi: 10.1016/j.annemergmed.2021.09.424. Epub 2021 Sep 24. PMID 34742591
- [Background] Southeast Asia Infectious Disease Clinical Research Network. Causes and outcomes of sepsis in southeast Asia: a multinational multicentre cross-sectional study. Lancet Glob Health. 2017 Feb;5(2):e157-e167. doi: 10.1016/S2214-109X(17)30007-4. PMID 28104185
- [Background] Gu X, Zhou F, Wang Y, Fan G, Cao B. Respiratory viral sepsis: epidemiology, pathophysiology, diagnosis and treatment. Eur Respir Rev. 2020 Jul 21;29(157):200038. doi: 10.1183/16000617.0038-2020. Print 2020 Sep 30. PMID 32699026
- [Background] Davenport EE, Burnham KL, Radhakrishnan J, Humburg P, Hutton P, Mills TC, Rautanen A, Gordon AC, Garrard C, Hill AV, Hinds CJ, Knight JC. Genomic landscape of the individual host response and outcomes in sepsis: a prospective cohort study. Lancet Respir Med. 2016 Apr;4(4):259-71. doi: 10.1016/S2213-2600(16)00046-1. Epub 2016 Feb 23. PMID 26917434
- [Background] Su Y, Chen D, Yuan D, Lausted C, Choi J, Dai CL, Voillet V, Duvvuri VR, Scherler K, Troisch P, Baloni P, Qin G, Smith B, Kornilov SA, Rostomily C, Xu A, Li J, Dong S, Rothchild A, Zhou J, Murray K, Edmark R, Hong S, Heath JE, Earls J, Zhang R, Xie J, Li S, Roper R, Jones L, Zhou Y, Rowen L, Liu R, Mackay S, O'Mahony DS, Dale CR, Wallick JA, Algren HA, Zager MA; ISB-Swedish COVID19 Biobanking Unit; Wei W, Price ND, Huang S, Subramanian N, Wang K, Magis AT, Hadlock JJ, Hood L, Aderem A, Bluestone JA, Lanier LL, Greenberg PD, Gottardo R, Davis MM, Goldman JD, Heath JR. Multi-Omics Resolves a Sharp Disease-State Shift between Mild and Moderate COVID-19. Cell. 2020 Dec 10;183(6):1479-1495.e20. doi: 10.1016/j.cell.2020.10.037. Epub 2020 Oct 28. PMID 33171100
- [Background] Taylor JC, Martin HC, Lise S, Broxholme J, Cazier JB, Rimmer A, Kanapin A, Lunter G, Fiddy S, Allan C, Aricescu AR, Attar M, Babbs C, Becq J, Beeson D, Bento C, Bignell P, Blair E, Buckle VJ, Bull K, Cais O, Cario H, Chapel H, Copley RR, Cornall R, Craft J, Dahan K, Davenport EE, Dendrou C, Devuyst O, Fenwick AL, Flint J, Fugger L, Gilbert RD, Goriely A, Green A, Greger IH, Grocock R, Gruszczyk AV, Hastings R, Hatton E, Higgs D, Hill A, Holmes C, Howard M, Hughes L, Humburg P, Johnson D, Karpe F, Kingsbury Z, Kini U, Knight JC, Krohn J, Lamble S, Langman C, Lonie L, Luck J, McCarthy D, McGowan SJ, McMullin MF, Miller KA, Murray L, Nemeth AH, Nesbit MA, Nutt D, Ormondroyd E, Oturai AB, Pagnamenta A, Patel SY, Percy M, Petousi N, Piazza P, Piret SE, Polanco-Echeverry G, Popitsch N, Powrie F, Pugh C, Quek L, Robbins PA, Robson K, Russo A, Sahgal N, van Schouwenburg PA, Schuh A, Silverman E, Simmons A, Sorensen PS, Sweeney E, Taylor J, Thakker RV, Tomlinson I, Trebes A, Twigg SR, Uhlig HH, Vyas P, Vyse T, Wall SA, Watkins H, Whyte MP, Witty L, Wright B, Yau C, Buck D, Humphray S, Ratcliffe PJ, Bell JI, Wilkie AO, Bentley D, Donnelly P, McVean G. Factors influencing success of clinical genome sequencing across a broad spectrum of disorders. Nat Genet. 2015 Jul;47(7):717-726. doi: 10.1038/ng.3304. Epub 2015 May 18. PMID 25985138
- [Background] Rautanen A, Mills TC, Gordon AC, Hutton P, Steffens M, Nuamah R, Chiche JD, Parks T, Chapman SJ, Davenport EE, Elliott KS, Bion J, Lichtner P, Meitinger T, Wienker TF, Caulfield MJ, Mein C, Bloos F, Bobek I, Cotogni P, Sramek V, Sarapuu S, Kobilay M, Ranieri VM, Rello J, Sirgo G, Weiss YG, Russwurm S, Schneider EM, Reinhart K, Holloway PA, Knight JC, Garrard CS, Russell JA, Walley KR, Stuber F, Hill AV, Hinds CJ; ESICM/ECCRN GenOSept Investigators. Genome-wide association study of survival from sepsis due to pneumonia: an observational cohort study. Lancet Respir Med. 2015 Jan;3(1):53-60. doi: 10.1016/S2213-2600(14)70290-5. Epub 2014 Dec 18. PMID 25533491
- [Background] Davenport EE, Antrobus RD, Lillie PJ, Gilbert S, Knight JC. Transcriptomic profiling facilitates classification of response to influenza challenge. J Mol Med (Berl). 2015 Jan;93(1):105-14. doi: 10.1007/s00109-014-1212-8. Epub 2014 Oct 28. PMID 25345603
- [Background] Dissanayake TK, Schauble S, Mirhakkak MH, Wu WL, Ng AC, Yip CCY, Lopez AG, Wolf T, Yeung ML, Chan KH, Yuen KY, Panagiotou G, To KK. Comparative Transcriptomic Analysis of Rhinovirus and Influenza Virus Infection. Front Microbiol. 2020 Jul 21;11:1580. doi: 10.3389/fmicb.2020.01580. eCollection 2020. PMID 32849329
- [Background] To KKW, Lu L, Fong CHY, Wu AKL, Mok KY, Yip CCY, Ke YH, Sze KH, Lau SKP, Hung IFN, Yuen KY. Rhinovirus respiratory tract infection in hospitalized adult patients is associated with TH2 response irrespective of asthma. J Infect. 2018 May;76(5):465-474. doi: 10.1016/j.jinf.2018.02.005. Epub 2018 Feb 15. PMID 29454786
- [Background] Khaliq W, Grossmann P, Neugebauer S, Kleyman A, Domizi R, Calcinaro S, Brealey D, Graler M, Kiehntopf M, Schauble S, Singer M, Panagiotou G, Bauer M. Lipid metabolic signatures deviate in sepsis survivors compared to non-survivors. Comput Struct Biotechnol J. 2020 Nov 21;18:3678-3691. doi: 10.1016/j.csbj.2020.11.009. eCollection 2020. PMID 33304464
- [Background] Wainberg M, Sinnott-Armstrong N, Mancuso N, Barbeira AN, Knowles DA, Golan D, Ermel R, Ruusalepp A, Quertermous T, Hao K, Bjorkegren JLM, Im HK, Pasaniuc B, Rivas MA, Kundaje A. Opportunities and challenges for transcriptome-wide association studies. Nat Genet. 2019 Apr;51(4):592-599. doi: 10.1038/s41588-019-0385-z. Epub 2019 Mar 29. PMID 30926968
- [Background] WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis. 2020 Aug;20(8):e192-e197. doi: 10.1016/S1473-3099(20)30483-7. Epub 2020 Jun 12. PMID 32539990
- [Background] GTEx Consortium. Human genomics. The Genotype-Tissue Expression (GTEx) pilot analysis: multitissue gene regulation in humans. Science. 2015 May 8;348(6235):648-60. doi: 10.1126/science.1262110. Epub 2015 May 7. PMID 25954001
- [Background] Tam V, Patel N, Turcotte M, Bosse Y, Pare G, Meyre D. Benefits and limitations of genome-wide association studies. Nat Rev Genet. 2019 Aug;20(8):467-484. doi: 10.1038/s41576-019-0127-1. PMID 31068683
- [Background] Howey R, Shin SY, Relton C, Davey Smith G, Cordell HJ. Bayesian network analysis incorporating genetic anchors complements conventional Mendelian randomization approaches for exploratory analysis of causal relationships in complex data. PLoS Genet. 2020 Mar 2;16(3):e1008198. doi: 10.1371/journal.pgen.1008198. eCollection 2020 Mar. PMID 32119656
- [Background] Davies NM, Holmes MV, Davey Smith G. Reading Mendelian randomisation studies: a guide, glossary, and checklist for clinicians. BMJ. 2018 Jul 12;362:k601. doi: 10.1136/bmj.k601. PMID 30002074
- [Background] Roadmap Epigenomics Consortium; Kundaje A, Meuleman W, Ernst J, Bilenky M, Yen A, Heravi-Moussavi A, Kheradpour P, Zhang Z, Wang J, Ziller MJ, Amin V, Whitaker JW, Schultz MD, Ward LD, Sarkar A, Quon G, Sandstrom RS, Eaton ML, Wu YC, Pfenning AR, Wang X, Claussnitzer M, Liu Y, Coarfa C, Harris RA, Shoresh N, Epstein CB, Gjoneska E, Leung D, Xie W, Hawkins RD, Lister R, Hong C, Gascard P, Mungall AJ, Moore R, Chuah E, Tam A, Canfield TK, Hansen RS, Kaul R, Sabo PJ, Bansal MS, Carles A, Dixon JR, Farh KH, Feizi S, Karlic R, Kim AR, Kulkarni A, Li D, Lowdon R, Elliott G, Mercer TR, Neph SJ, Onuchic V, Polak P, Rajagopal N, Ray P, Sallari RC, Siebenthall KT, Sinnott-Armstrong NA, Stevens M, Thurman RE, Wu J, Zhang B, Zhou X, Beaudet AE, Boyer LA, De Jager PL, Farnham PJ, Fisher SJ, Haussler D, Jones SJ, Li W, Marra MA, McManus MT, Sunyaev S, Thomson JA, Tlsty TD, Tsai LH, Wang W, Waterland RA, Zhang MQ, Chadwick LH, Bernstein BE, Costello JF, Ecker JR, Hirst M, Meissner A, Milosavljevic A, Ren B, Stamatoyannopoulos JA, Wang T, Kellis M. Integrative analysis of 111 reference human epigenomes. Nature. 2015 Feb 19;518(7539):317-30. doi: 10.1038/nature14248. PMID 25693563
- [Background] Yang JK, Wang YY, Liu C, Shi TT, Lu J, Cao X, Yang FY, Feng JP, Chen C, Ji LN, Xu A. Urine Proteome Specific for Eye Damage Can Predict Kidney Damage in Patients With Type 2 Diabetes: A Case-Control and a 5.3-Year Prospective Cohort Study. Diabetes Care. 2017 Feb;40(2):253-260. doi: 10.2337/dc16-1529. Epub 2016 Nov 30. PMID 27903615
- [Background] Harati MD, Williams RR, Movassaghi M, Hojat A, Lucey GM, Yong WH. An Introduction to Starting a Biobank. Methods Mol Biol. 2019;1897:7-16. doi: 10.1007/978-1-4939-8935-5_2. PMID 30539430
- [Background] Jain S, Self WH, Wunderink RG, Fakhran S, Balk R, Bramley AM, Reed C, Grijalva CG, Anderson EJ, Courtney DM, Chappell JD, Qi C, Hart EM, Carroll F, Trabue C, Donnelly HK, Williams DJ, Zhu Y, Arnold SR, Ampofo K, Waterer GW, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, McCullers JA, Pavia AT, Edwards KM, Finelli L; CDC EPIC Study Team. Community-Acquired Pneumonia Requiring Hospitalization among U.S. Adults. N Engl J Med. 2015 Jul 30;373(5):415-27. doi: 10.1056/NEJMoa1500245. Epub 2015 Jul 14. PMID 26172429
- [Background] Niederman MS, Mandell LA, Anzueto A, Bass JB, Broughton WA, Campbell GD, Dean N, File T, Fine MJ, Gross PA, Martinez F, Marrie TJ, Plouffe JF, Ramirez J, Sarosi GA, Torres A, Wilson R, Yu VL; American Thoracic Society. Guidelines for the management of adults with community-acquired pneumonia. Diagnosis, assessment of severity, antimicrobial therapy, and prevention. Am J Respir Crit Care Med. 2001 Jun;163(7):1730-54. doi: 10.1164/ajrccm.163.7.at1010. No abstract available. PMID 11401897
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Field N, Cohen T, Struelens MJ, Palm D, Cookson B, Glynn JR, Gallo V, Ramsay M, Sonnenberg P, Maccannell D, Charlett A, Egger M, Green J, Vineis P, Abubakar I. Strengthening the Reporting of Molecular Epidemiology for Infectious Diseases (STROME-ID): an extension of the STROBE statement. Lancet Infect Dis. 2014 Apr;14(4):341-52. doi: 10.1016/S1473-3099(13)70324-4. Epub 2014 Mar 14. PMID 24631223
- [Background] Cohen JF, Korevaar DA, Altman DG, Bruns DE, Gatsonis CA, Hooft L, Irwig L, Levine D, Reitsma JB, de Vet HC, Bossuyt PM. STARD 2015 guidelines for reporting diagnostic accuracy studies: explanation and elaboration. BMJ Open. 2016 Nov 14;6(11):e012799. doi: 10.1136/bmjopen-2016-012799. PMID 28137831
- See also: The Human Protein Atlas. Accessed 15th September 2021 — https://www.proteinatlas.org
- See also: Hall A. Eight things you should consider before setting up a biobank. Human Tissue Authority. Accessed on 15th September 2021 — https://www.hta.gov.uk/blog/eight-things-you-should-consider-setting-biobank
- See also: Accessed on 22nd July 2021 — https://www.strobe-statement.org/index.php?id=available-checklists
- See also: Accessed on 22nd July 2021 — https://www.equator-network.org/reporting-guidelines/tripod-statement/
- See also: Coronavirus (COVID-19). Accessed 16th September 2021 — https://news.google.com/covid19/map?hl=en-GB&gl=GB&ceid=GB%3Aen